CLINICAL TRIAL: NCT00703248
Title: The Human Immunodeficiency Virus and Osteopathic Manipulation Evaluation Study
Acronym: HOME
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Southeastern University (Other)
Responsible Party: Mark A Newberry
Purpose: Supportive Care
Other Study IDs: HPD-OST10030701
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2008-07-08 (Estimated); Status verified 2008-06

CONDITIONS: HIV Infections
Keywords: Human Immunodeficiency Virus (HIV); complementary therapies
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Manipulation, Osteopathic

ARMS (2):
- 1 (Experimental)
  Interventions: Procedure: Osteopathic Manipulative Treatments
- 2 (No Intervention)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatments — 1. opening the thoracic inlet
  2. pectoral traction for 1 minute bilaterally
  3. rib raising for a total of 4 minutes- 2 minutes on each side of the thoracic spine ]
  4. thoracic pump at a rate of 60 times per minute for a total of 5 minutes bilaterally
  5. abdominal pump at a rate of 30 times per minute for a total of 5 minutes bilaterally.
  Arms: 1

SUMMARY:
Treatment options that increase immune function, such as Osteopathic Manipulation Treatment (OMT) lymphatic techniques, may provide improved short or long term performance of the immune system. However, the efficacy of OMT to boost immune function among people living with HIV has not yet been examined in a controlled study. Our experiment is designed to examine the short (45 minutes) term impact of OMT on the white blood cells counts of HIV positive men who are either antiretroviral therapy (ART) naïve or have not taken ART for at least 12 months prior to enrollment in the study.

ELIGIBILITY:
Inclusion Criteria:

* are either Antiretroviral Therapy (ART) naïve or not have taken ART for the past 12 months
* are between the ages of 18 to 65
* have a CD4+ T cell count between 200-700cells/mm3
* have viral loads less than 100,000 copies/mL
* do not have any medical condition that limits his ability to participate in this study as defined by his physician (e.g., cancer, blood clotting disorder etc.)
* are willing to provide informed consent
* are not using any drugs recreationally
* are not on prescribed systemic steroids
* are willing to recruit a friend/partner, aware of the their HIV serostatus, to be trained in OMT techniques and apply it to him daily.

Exclusion Criteria:

* history of malignancy excluding both squamous cell carcinoma and basal cell carcinoma of the skin and/or any malignancies fully treated and considered cured by the treating physician for at least 1 year
* aortic aneurism/disease
* vertebral artery disease
* carotid artery stenosis/disease
* abdominal hernias
* portal hypertension
* cirrhosis
* cervical disc disease currently exhibiting radicular symptomatology (i.e. numbness, burning, muscle weakness, etc)
* infectious mononucleosis in the past 12 weeks,
* pneumothorax
* bone disease
* Participants with a medical access port and/or a noncompliant ribcage will be excluded from the study.
* The potential causes for ribcage noncompliance include:

  * congestive obstructive pulmonary disorder (COPD)
  * spinal arthritis
  * costochondritis
  * congestive heart failure (CHF)
  * pulmonary edema
  * recent trauma to the ribcage
  * certain connective tissue disease such as Ankylosing Spondylitis
* There is a risk of abdominal aortic aneurysm (AAA) rupture in participants with AAA and these participants are excluded from the study.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2007-10; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States